CLINICAL TRIAL: NCT02723591
Title: Astagraf XL® to Understand the Impact of Immunosuppression on De Novo DSA Development and Chronic Immune Activation in Kidney Transplantation
Brief Title: To Compare the Effects of Immediate-release Tacrolimus and Astagraf XL on Donor-Specific Antibody (DSA) Formation and the Development of Immune Activation (IA) in de Novo Kidney Transplant Recipients
Acronym: ASTOUND
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IDTX-MA-3004; 2018-003867-79 (EudraCT Number)
Record Dates: First submitted 2016-03-03; First posted 2016-03-30 (Estimated); Results first posted 2020-06-29 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-11

CONDITIONS: Kidney Transplantation
Keywords: FK506; Kidney Transplantation; Tacrolimus; Astagraf XL
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tacrolimus, Extended Release (Astagraf XL®) Once Daily (Active Comparator): Participants received tacrolimus extended release (Astagraf XL) at a starting dose of 0.15 milligram per kilogram (mg/kg), once daily, orally within 48 hours of transplantation (per the treating physician's discretion) for up to 1 year. Dose adjustments were allowed such that participants receiving tacrolimus maintained a minimal trough concentration of 6 nanogram per milliliter (ng/mL) at all times during the study.
  Interventions: Drug: Tacrolimus
- Tacrolimus, Immediate Release Twice Daily (BID) (Active Comparator): Participants received tacrolimus immediate release as per the institutionally-derived protocol, BID, orally within 48 hours of transplantation (per the treating physician's discretion) for up to 1 year. Dose adjustments were allowed such that participants receiving tacrolimus maintained a minimal trough concentration of 6 ng/mL at all times during the study.
  Interventions: Drug: Tacrolimus immediate release

INTERVENTIONS:
Drug: Tacrolimus — Oral Capsule
  Other Names: Advagraf; FK506E; Astagraf XL
  Arms: Tacrolimus, Extended Release (Astagraf XL®) Once Daily
Drug: Tacrolimus immediate release — Oral Capsule
  Other Names: FK506; Prograf; generic immediate release tacrolimus
  Arms: Tacrolimus, Immediate Release Twice Daily (BID)

SUMMARY:
This study compared the incidence of a two-part composite endpoint consisting of de novo donor specific antibody (DSA) formation or a designation of immune activation (IA) on peripheral blood molecular profiling in participants maintained on twice daily, immediate-release tacrolimus versus those maintained on Astagraf XL in the first year post-transplant.

DETAILED DESCRIPTION:
This was an exploratory, two year (shortened to 1 year due to a stopping rule necessitated by the adaptive design), prospective, randomized, multi-center, open-label trial examining long-term kidney transplant outcomes through the use of an adaptive design and a two-part, composite surrogate endpoint. Specifically, it was designed to compare the effects of twice daily, immediate-release tacrolimus and once daily Astagraf XL on DSA formation and the development of a peripheral blood molecular profile indicating the presence of IA in de novo kidney transplant recipients during the first year following transplantation. For the purposes of this study, IA was defined as a positive molecular signature using a molecular assay in all participants.

Participants were screened prior to surgery and randomized 1:1 to receive immediate-release tacrolimus, administered twice daily, or Astagraf XL, as a component of a standard immunosuppression maintenance regimen also consisting of corticosteroids (if given per institutional protocol) and mycophenolate mofetil (MMF) (or Myfortic® equivalent). Investigators were encouraged to start participants on the randomized study treatment (immediate release tacrolimus or Astagraf XL) within 48 hours of transplantation (pre-transplant administration of study treatment was not allowed). However, if medically indicated per the treating physician's discretion, initiation of study treatment was delayed for up to seven days post-transplant.

ELIGIBILITY:
Inclusion Criteria:

* Recipient of a de novo kidney from a living or deceased donor. Note: Recipient of an en bloc deceased donor kidney transplant from a pediatric donor ≥5 years of age AND weighing greater than 20 kg is allowed.
* If deceased donor, a Kidney Donor Profile Index (KDPI) ≤ 85 (Donation after Circulatory Death [DCD] and what was previously known as extended criteria donor [ECD] organ recipients are eligible for enrollment provided KDPI ≤85).
* At least one antigen mismatch at major Major Histocompatibility Complex (MHC) (class I or class II).
* Willingness to comply with study protocol.
* Subject agrees not to participate in another investigational drug study while on treatment.
* Female subject must be either:

  a. Of non-child-bearing potential i. Post-menopausal (defined as at least 1 year without any menses) prior to screening, or ii. Documented surgically sterile or status post-hysterectomy b. Or, if of childbearing potential, i. Agree not to try to become pregnant during the study and for 90 days after the final study drug administration ii. And have a negative serum or urine pregnancy test within 7 days prior to transplant procedure iii. And, if heterosexually active, agree to consistently use two forms of highly effective birth control (at least one of which must be a barrier method) which includes consistent and correct usage of established oral contraception, established intrauterine device or intrauterine system, or barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository or vasectomy in the male partner, starting at screening and throughout the study period and for 90 days after the final study drug administration.
* Male subject and their female spouse/partners who are of childbearing potential must be using highly effective contraception consisting of two forms of birth control (one of which must be a barrier method) starting at screening and continuing throughout the study period and for 90 days after the final study drug administration.
* Male subject must not donate sperm starting at screening throughout the study period and for 90 days after the final study drug administration.
* Female subject must agree not to breastfeed starting at screening and throughout the study period, and for 90 days after the final study drug administration.
* Female subject must not donate ova starting at screening and throughout the study period, and for 90 days after the final study drug administration.
* Will be receiving induction immunotherapy (either T-cell depleting agent, anti-CD52 monoclonal antibody, or Interleukin-2 (IL-2) co-stimulation blocker), with dose and frequency of the chosen induction agent determined by local standard of care. Steroid-only induction therapy does not satisfy this criterion.

Exclusion Criteria:

* Patient is known to have a positive test for latent Tuberculosis (TB) and has not previously received adequate anti-microbial therapy or would require TB prophylaxis after transplant.
* Uncontrolled concomitant infection or any unstable medical condition that could interfere with study objectives.
* Significant liver disease, defined as having, during the past 28 days, consistently elevated Aspartate Aminotransferase, GOT (AST) Serum Glutamic Oxaloacetic Transaminase (SGOT) and/or Alanine Aminotransferase, GPT (ALT) Serum Glutamic Pyruvic Transaminase (SPGT) levels greater than 3 times the upper value of the normal range of the investigational site.
* Patient currently taking or maintained on another form of extended-release tacrolimus following his/her transplant procedure.
* Patient who will be maintained on a non-tacrolimus-based maintenance immunosuppressive regimen following his/her transplant procedure.
* Patient currently taking, having taken within 30 days, or who will be maintained on an Mammalian target of rapamycin (mTOR) inhibitor following his/her transplant procedure.
* Use of an investigational study drug in the 30 days prior to the transplant procedure.
* Contraindication or hypersensitivity to drugs or any of their components that constitute the immunosuppression regimen.
* 6 Antigen (Ag) match or zero mismatch at major Major Histocompatibility Complex (MHC) (class I or class II).
* Receipt of an Blood Group System (A, B, AB, and O) (ABO)-incompatible organ. Note: A2 donor to O recipient or A2 donor to B recipient is considered ABO-compatible and not excluded by this criterion.
* Presence of current or historic pre-formed anti-Human Leukocyte Antigen (HLA) DSA against the current donor (evidence of pre-formed, non-donor HLA is not exclusionary) as defined by a subject meeting any of the following criteria*: a) positive virtual crossmatch, b) positive T- or B-cell crossmatch by National Institutes of Health (NIH) antiglobulin lymphocytotoxicity method** , c) .Positive T- or B-cell flow cytometry crossmatch defined by the Multiparameter flow cytometry (MFC) criteria used by the center's HLA lab for their local proficiency testing.,** d) An Mean Fluorescence Intensity (MFI) greater than or approaching 1000 using flow cytometry/Luminex-based, specific anti-HLA antibody testing.

  * * Patients are eligible to enroll with a negative virtual crossmatch if used in lieu of a physical crossmatch, if, use of such is required to obviate the accrual of excessive ischemia time. However, continued participation is predicated on the performance of the physical crossmatch within 48 hours of transplant. If the physical crossmatch is positive, the subject will be discontinued.
  * ** If b or c above are positive secondary to a suspected positive auto-crossmatch, that is not exclusionary as long as a and b above are not met.
* Receipt of desensitization, antibody-removal, anti-B-cell, or anti-plasma cell therapy in the 90 days preceding the transplant procedure.
* Planned initiation (prior to transplant) of desensitization, antibody-removal, anti-B-cell, or anti-plasma cell therapy within 7 days of the transplant procedure.
* Donor or recipient with known hepatitis C infection (Hepatitis C Virus (HCV) antibody positive), Human Immunodeficiency Virus (HIV) infection (HIV antibody positive), acute hepatitis B infection (Hepatitis B Surface Antigen (HBsAg) positive, anti-Hepatitis B Virus Core (HBc) positive, Immunoglobulin M (IgM) anti-HBc positive, anti-HBs negative) chronic hepatitis B infection (HBsAg positive, anti-HBc positive, IgM anti-HBc negative, anti-HBs negative), or equivocal hepatitis B status (HBsAg negative, anti-HBc positive, anti-HBs negative). Patients (donor or recipient) who have normal liver function tests (LFT) and who are either hepatitis C positive with a negative viral load or have natural or vaccine-acquired immunity from hepatitis B are not excluded by this criterion.
* Primary focal segmental glomerulosclerosis.
* Subject has a current malignancy or history of malignancy (within the past 5 years), except non-metastatic basal or squamous cell carcinoma of the skin or carcinoma-in-situ of the cervix that has been successfully treated.
* Recipient of multi-organ or dual kidney transplants (inclusive of current transplant and any prior non-renal transplants). Note: Patients with prior kidney transplants are eligible.
* Recipient of an en bloc, pediatric deceased donor kidney from a donor less than 5 years of age OR weighing less than 20 kg.
* Prior graft loss secondary to Cytomegalovirus (CMV) or BK nephropathy.
* Prior history of invasive organ disease in the presence of CMV or BKV or clinically significant CMV viremia.
* History of clinically significant BK viruria.
* Any condition which makes the subject unsuitable for study participation.
* Planned complete steroid avoidance (Steroid initiation and subsequent taper / withdrawal will be allowed and will be under the purview of the treating physician).
* Planned receipt of post-transplant prophylactic HCV treatment.

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 599 (Actual)
Dates: Start 2016-09-09 (Actual); Primary Completion 2019-06-14 (Actual); Study Completion 2019-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Astellas Medical Affairs, Americas
Locations (30):
- United States (30):
  - Site US10006, Birmingham, Alabama
  - Site US10025, Scottsdale, Arizona
  - Site US10031, Los Angeles, California
  - Site US10005, Sacramento, California
  - Site US10016, San Francisco, California
  - Site US10024, Aurora, Colorado
  - Site US10003, New Haven, Connecticut
  - Site US10014, Washington D.C., District of Columbia
  - Site US10030, Jacksonville, Florida
  - Site US10020, Chicago, Illinois
  - Site US10010, Chicago, Illinois
  - Site US10001, Baltimore, Maryland
  - Site US10007, Boston, Massachusetts
  - Site US10013, Ann Arbor, Michigan
  - Site US10032, Detroit, Michigan
  - Site US10029, Minneapolis, Minnesota
  - Site US10027, Rochester, Minnesota
  - Site US10019, Livingston, New Jersey
  - Site US10004, Buffalo, New York
  - Site US10037, New York, New York
  - Site US10022, New York, New York
  - Site US10028, New York, New York
  - Site US10021, Syracuse, New York
  - Site US10026, Portland, Oregon
  - Site US10002, Charleston, South Carolina
  - Site US10036, Houston, Texas
  - Site US10018, Salt Lake City, Utah
  - Site US10012, Charlottesville, Virginia
  - Site US10008, Falls Church, Virginia
  - Site US10023, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- See also: Link to results on the Astellas Clinical Study Results website. — https://astellasclinicalstudyresults.com/study.aspx?ID=375

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants of ≥16 years and ≤70 of age requiring kidney transplant were enrolled. Randomization was stratified by alemtuzumab (yes/no), kidney donor profile index (KDPI) (3 levels: N/A [living donors] versus ≤50 versus >50), and human leukocyte antigens (HLA) Class II mismatch (yes/no).
Groups:
- Tacrolimus, Extended Release (Astagraf XL®) Once Daily: Participants received tacrolimus extended release capsule (Astagraf XL) at a starting dose of 0.15 milligram per kilogram (mg/kg), once daily, orally within 48 hours of transplantation (per the treating physician's discretion) for up to 1 year. Dose adjustments were allowed such that participants receiving tacrolimus maintained a minimal trough concentration of 6 nanogram per milliliter (ng/mL) at all times during the study.
- Tacrolimus, Immediate Release Twice Daily (BID): Participants received tacrolimus immediate release capsule as per the institutionally-derived protocol, BID, orally within 48 hours of transplantation (per the treating physician's discretion) for up to 1 year. Dose adjustments were allowed such that participants receiving tacrolimus maintained a minimal trough concentration of 6 ng/mL at all times during the study.
Period: Overall Study
Arm/Group | Tacrolimus, Extended Release (Astagraf XL®) Once Daily | Tacrolimus, Immediate Release Twice Daily (BID)
Started | 300 | 299
Completed | 204 | 198
Not Completed | 96 | 101
Not completed — Adverse Event | 48 | 40
Not completed — Death | 2 | 2
Not completed — Lack of Efficacy | 4 | 3
Not completed — Lost to Follow-up | 1 | 7
Not completed — Protocol Violation | 20 | 23
Not completed — Withdrawal by Subject | 4 | 8
Not completed — Randomized but Never Received StudyDrug | 12 | 12
Not completed — Miscellaneous | 5 | 6

BASELINE CHARACTERISTICS:
Population: The randomized set consisted of all participants who were randomized to receive the study drug (Astagraf XL or BID tacrolimus).
Groups:
- Tacrolimus, Extended Release (Astagraf XL®) Once Daily: Participants received tacrolimus extended release capsule (Astagraf XL) at a starting dose of 0.15 mg/kg, once daily, orally within 48 hours of transplantation (per the treating physician's discretion) for up to 1 year. Dose adjustments were allowed such that participants receiving tacrolimus maintained a minimal trough concentration of 6 ng/mL at all times during the study.
- Tacrolimus, Immediate Release BID: Participants received tacrolimus immediate release capsule as per the institutionally-derived protocol, BID, orally within 48 hours of transplantation (per the treating physician's discretion) for up to 1 year. Dose adjustments were allowed such that participants receiving tacrolimus maintained a minimal trough concentration of 6 ng/mL at all times during the study.
- Total: Total of all reporting groups
Arm/Group | Tacrolimus, Extended Release (Astagraf XL®) Once Daily | Tacrolimus, Immediate Release BID | Total
Number analyzed (Participants) | 300 | 299 | 599
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49 (11.7) | 48.5 (11.6) | 48.8 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 111 | 91 | 202
  Male | 189 | 208 | 397
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 32 | 34 | 66
  Not Hispanic or Latino | 268 | 265 | 533
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 1 | 5
  Asian | 10 | 14 | 24
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 3
  Black or African American | 58 | 67 | 125
  White | 212 | 200 | 412
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 14 | 16 | 30

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Were Positive for de Novo DSA (dnDSA) or Immune Activation (IA) Occurrence
Description: DSA was considered as a categorical (binary) variable with positivity determined at a threshold criteria approaching mean fluorescence intensity (MFI)=1000 at any time during the study. IA was considered either present or absent using the Trugraf™ v2.0 molecular assay. A negative designation (Trugraf TX Normal) was referred to as Immune Quiescence (IQ). Due to operating characteristics of the assay, a positive designation was considered evidence of IA in all participants.
Time Frame: From date of transplant until 1 year
Population: The Modified Full Analysis Set (mFAS) consisted of all participants who were randomized and who received at least 1 dose of study drug (Astagraf XL or BID tacrolimus), and whose pretransplant cross-matched antibody samples did not demonstrate preformed DSA for the duration of the study.
Measure: Number; unit: percentage of participants
Arm/Group | Tacrolimus, Extended Release (Astagraf XL®) Once Daily | Tacrolimus, Immediate Release BID
Number analyzed (Participants) | 275 | 279
percentage of participants | 35.6 | 34.4
Statistical Analysis 1: Comparison: Tacrolimus, Extended Release (Astagraf XL®) Once Daily vs Tacrolimus, Immediate Release BID; Logistic regression with DSA/IA occurrence by Month 12 as response, with treatment group, planned Campath use, KDPI level (as recorded in IVRS), HLA Class II mismatch, recipient age, recipient gender, recipient race, and pre-transplant calculated panel reactivity antibody (cPRA) as fixed effects, and pooled site as a random effect with standard variance components covariance type; Test type: Superiority; p = 0.5777, Regression, Logistic; Odds Ratio (OR) = 1.115, 95% CI 2-sided [0.760 to 1.636]

2. Secondary Outcome: Percentage of Participants Who Were Positive, Negative or Indeterminate for dnDSA Occurrence
Description: DSA was considered as a categorical (binary) variable with positivity determined at a threshold criteria approaching MFI=1000 at any time during the study. Indeterminate was defined as MFI signal was >1000 and DSA was suspected, but could not be confirmed due to inadequate donor typing. Participants whose samples for the test were not available were reported as unknown.
Time Frame: From date of transplant until 1 year
Population: The mFAS consisted of all participants who were randomized and who received at least 1 dose of study drug (Astagraf XL or BID tacrolimus), and whose pretransplant cross-matched antibody samples did not demonstrate preformed DSA for the duration of the study.
Measure: Number; unit: percentage of participants
Arm/Group | Tacrolimus, Extended Release (Astagraf XL®) Once Daily | Tacrolimus, Immediate Release BID
Number analyzed (Participants) | 275 | 279
percentage of participants
  Positive | 5.5 | 4.3
  Negative | 90.5 | 92.8
  Indeterminate | 4 | 2.5
  Unknown | 0 | 0.4

3. Secondary Outcome: Peak Mean Fluorescence Intensity (MFI) of DSA Positive Participants
Description: Peak MFI of DSA positive participants was reported.
Time Frame: From date of transplant until 1 year
Population: The mFAS consisted of all participants who were randomized and who received at least 1 dose of study drug (Astagraf XL or BID tacrolimus), and whose pretransplant cross-matched antibody samples did not demonstrate preformed DSA for the duration of the study. Only those mFAS participants who tested positive for dnDSA were included in the analyses.
Measure: Median (Full Range); unit: fluorescence intensity unit
Arm/Group | Tacrolimus, Extended Release (Astagraf XL®) Once Daily | Tacrolimus, Immediate Release BID
Number analyzed (Participants) | 15 | 12
fluorescence intensity unit | 6119.21 [1320.0 to 29317.6] | 2727.99 [1066.0 to 19971.5]

4. Secondary Outcome: Percentage of DSA Positive Participants With Weak, Moderate and Strong Antibody Strentgh
Description: DSA was considered as a categorical (binary) variable with positivity determined at a threshold criteria approaching MFI=1000 at any time during the study.
Time Frame: From date of transplant until 1 year
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Tacrolimus, Extended Release (Astagraf XL®) Once Daily | Tacrolimus, Immediate Release BID
Number analyzed (Participants) | 15 | 12
percentage of participants
  Weak | 0 | 0
  Moderate | 73.3 | 83.3
  Strong | 26.7 | 16.7
Statistical Analysis 1: Comparison: Tacrolimus, Extended Release (Astagraf XL®) Once Daily vs Tacrolimus, Immediate Release BID; P-values obtained from a 2x3 Exact Test of treatment by strength levels; Test type: Superiority; p = 0.6618, Fisher Exact

5. Secondary Outcome: Percentage of DSA Positive Participants With DSA Persistence
Description: DSA was regarded as persistent under the following conditions: (i) DSA was detected and remained above the threshold for positivity (MFI = 1000) for two consecutive or nonconsecutive measurements, or (ii) the new appearance of a DSA at the threshold for positivity when preceded by a DSA of a different specificity that had subsequently become non-detectable.
Time Frame: From date of transplant until 1 year
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Tacrolimus, Extended Release (Astagraf XL®) Once Daily | Tacrolimus, Immediate Release BID
Number analyzed (Participants) | 15 | 12
percentage of participants | 73.3 | 50

6. Secondary Outcome: Percentage of Participants Who Were Positive or Negative for Complement Component 1, Q Subcomponent (C1q)-Binding DSA
Description: Percentage of participants who were positive or negative for C1q-binding DSA were reported.
Time Frame: From date of transplant until 1 year
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Tacrolimus, Extended Release (Astagraf XL®) Once Daily | Tacrolimus, Immediate Release BID
Number analyzed (Participants) | 275 | 279
percentage of participants
  Positive | 1.8 | 0.4
  Negative | 98.2 | 99.6

7. Secondary Outcome: Percentage of Participants Who Were Positive or Negative for DSA Immunoglobulin G (IgG3) Isotype
Description: Percentage of participants who were positive or negative for IgG3 isotype were reported.
Time Frame: From date of transplant until 1 year
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Tacrolimus, Extended Release (Astagraf XL®) Once Daily | Tacrolimus, Immediate Release BID
Number analyzed (Participants) | 275 | 279
percentage of participants
  Positive | 0.7 | 1.1
  Negative | 99.3 | 98.9

8. Secondary Outcome: Percentage of DSA Positive Participants With Human Leukocyte Antigen, Class II, DQ Locus (HLA-DQ)
Description: Percentage of DSA positive participants with HLA-DQ Class-II were reported.
Time Frame: From date of transplant until 1 year
Population: The mFAS consisted of all participants who were randomized and who received at least 1 dose of study drug (Astagraf XL or BID tacrolimus), and whose pretransplant cross-matched antibody samples did not demonstrate preformed DSA for the duration of the study. Only those mFAS participants who tested positive for DSA were included in the analyses.
Measure: Number; unit: percentage of participants
Arm/Group | Tacrolimus, Extended Release (Astagraf XL®) Once Daily | Tacrolimus, Immediate Release BID
Number analyzed (Participants) | 15 | 12
percentage of participants | 40 | 25

9. Secondary Outcome: Percentage of Participants Who Were Positive for IA Occurrence From Day 1 to Day 365 Visit
Description: IA was considered either present or absent using the Trugraf™ v2.0 molecular assay. A negative designation (Trugraf TX Normal) was referred to as Immune Quiescence (IQ). Due to operating characteristics of the assay, a positive designation was considered evidence of IA in all participants.
Time Frame: From day 1 to day 365 visit
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Tacrolimus, Extended Release (Astagraf XL®) Once Daily | Tacrolimus, Immediate Release BID
Number analyzed (Participants) | 275 | 279
percentage of participants | 31.3 | 31.2
Statistical Analysis 1: Comparison: Tacrolimus, Extended Release (Astagraf XL®) Once Daily vs Tacrolimus, Immediate Release BID; Logistic regression with IA occurrence by Month 12 as response, with treatment group, planned Campath use, KDPI level (as recorded in IVRS), HLA Class II mismatch, recipient age, recipient gender, recipient race, and pre-transplant cPRA as fixed effects, and pooled site as a random effect with standard Variance Components covariance type; Test type: Superiority; p = 0.8518, Regression, Logistic; Odds Ratio (OR) = 1.038, 95% CI 2-sided [0.700 to 1.539]

10. Secondary Outcome: Percentage of Participants Who Were Positive for IA Occurrence From Day 30 to Day 365 Visit
Description: as for outcome 9
Time Frame: From day 30 to day 365 visit
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Tacrolimus, Extended Release (Astagraf XL®) Once Daily | Tacrolimus, Immediate Release BID
Number analyzed (Participants) | 275 | 279
percentage of participants | 21.8 | 21.9

11. Secondary Outcome: Percentage of Participants With IA Persistence
Description: IA was regarded as persistent under the following conditions: (i) IA was detected and remained above the threshold for positivity for two consecutive or non-consecutive measurements, or (ii) the new appearance of an IA at the threshold for positivity when preceded by an IA of a different specificity that had subsequently become non-detectable.
Time Frame: From date of transplant until 1 year
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Tacrolimus, Extended Release (Astagraf XL®) Once Daily | Tacrolimus, Immediate Release BID
Number analyzed (Participants) | 275 | 279
percentage of participants | 7.3 | 10

12. Secondary Outcome: Percentage of Participants With Presence of Transplant Glomerulopathy (TG) on Biopsy
Description: TG was defined as chronic glomerulopathy (cg) >0 on centrally-interpreted institutional protocol biopsy or biopsy obtained for cause during the first year post-transplant with +2 months visit window.
Time Frame: From date of transplant until month 14
Population: The Biopsy Analysis Dataset (BAS) consisted of all mFAS participants who had at least 1 post-transplant central pathology assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Tacrolimus, Extended Release (Astagraf XL®) Once Daily | Tacrolimus, Immediate Release BID
Number analyzed (Participants) | 123 | 136
percentage of participants | 6.5 | 6.6
Statistical Analysis 1: Comparison: Tacrolimus, Extended Release (Astagraf XL®) Once Daily vs Tacrolimus, Immediate Release BID; P-values obtained from a 2-sided Fisher's Exact Test of treatment arm by response; Test type: Superiority; p = 1.0000, Fisher Exact

13. Secondary Outcome: Percentage of Participants With Presence of Microcirculatory Inflammation (MI) on Biopsy
Description: MI was defined as glomerulitis (g) + peritubular capillaritis (ptc)>=2 on centrally-interpreted institutional protocol biopsy or biopsy obtained for cause during the first year post-transplant, with +2 months visit window.
Time Frame: From date of transplant until month 14
Population: The BAS consisted of all mFAS participants who had at least 1 post-transplant central pathology assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Tacrolimus, Extended Release (Astagraf XL®) Once Daily | Tacrolimus, Immediate Release BID
Number analyzed (Participants) | 123 | 136
percentage of participants | 8.9 | 5.9
Statistical Analysis 1: Comparison: Tacrolimus, Extended Release (Astagraf XL®) Once Daily vs Tacrolimus, Immediate Release BID; P-values obtained from a 2-sided Fisher's Exact Test of treatment arm by response; Test type: Superiority; p = 0.4750, Fisher Exact

14. Secondary Outcome: Percentage of Participants With Presence of Interstitial Fibrosis and Tubular Atrophy (IFTA) and Inflammation on Biopsy
Description: IFTA and inflammation was defined as IFTA positive and inflammation positive (i >0) on centrally-interpreted institutional protocol biopsy or biopsy obtained for cause during the first year posttransplant, with +2 months visit window.
Time Frame: From date of transplant until month 14
Population: The BAS consisted of all mFAS participants who had at least 1 post-transplant central pathology assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Tacrolimus, Extended Release (Astagraf XL®) Once Daily | Tacrolimus, Immediate Release BID
Number analyzed (Participants) | 123 | 136
percentage of participants | 26 | 16.9
Statistical Analysis 1: Comparison: Tacrolimus, Extended Release (Astagraf XL®) Once Daily vs Tacrolimus, Immediate Release BID; P-values obtained from a 2-sided Fisher's Exact Test of treatment arm by response; Test type: Superiority; p = 0.0939, Fisher Exact

15. Secondary Outcome: Percentage of Participants With Estimated Glomerular Filtration Rate (eGFR) Threshold of <30 Millimetre Per Minute Per 1.73 Meter Square (mL/Min/1.73m^2)
Description: The eGFR was calculated using the Modification of Diet in Renal Disease (MDRD) formula.
Time Frame: At 1 year post transplant
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Tacrolimus, Extended Release (Astagraf XL®) Once Daily | Tacrolimus, Immediate Release BID
Number analyzed (Participants) | 275 | 279
percentage of participants | 1.5 | 1.8

16. Secondary Outcome: Percentage of Participants With eGFR Threshold of <40 mL/Min/1.73m^2
Description: The eGFR was calculated using the MDRD formula.
Time Frame: At 1 year post transplant
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Tacrolimus, Extended Release (Astagraf XL®) Once Daily | Tacrolimus, Immediate Release BID
Number analyzed (Participants) | 275 | 279
percentage of participants | 9.5 | 5.7

17. Secondary Outcome: Percentage of Participants With eGFR Threshold of <50 mL/Min/1.73m^2
Description: The eGFR was calculated using the MDRD formula.
Time Frame: At 1 year post transplant
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Tacrolimus, Extended Release (Astagraf XL®) Once Daily | Tacrolimus, Immediate Release BID
Number analyzed (Participants) | 275 | 279
percentage of participants | 25.5 | 19.7
Statistical Analysis 1: Comparison: Tacrolimus, Extended Release (Astagraf XL®) Once Daily vs Tacrolimus, Immediate Release BID; Logistic regression with occurrence of eGFR < 50 by Month 12 as response, with treatment group, planned Campath use, KDPI level (as recorded in IVRS), HLA Class II mismatch, recipient age, recipient gender, recipient race, and pre-transplant cPRA as fixed effects, and pooled site as a random effect with standard Variance Components covariance type; Test type: Superiority; p = 0.1160, Regression, Logistic; Odds Ratio (OR) = 1.431, 95% CI 2-sided [0.915 to 2.240]

18. Secondary Outcome: Percentage of Participants With a Five-point Decline in eGFR
Description: The eGFR was calculated using the MDRD formula.
Time Frame: From 30 days post transplant until 1 year
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Tacrolimus, Extended Release (Astagraf XL®) Once Daily | Tacrolimus, Immediate Release BID
Number analyzed (Participants) | 275 | 279
percentage of participants | 13.1 | 11.1
Statistical Analysis 1: Comparison: Tacrolimus, Extended Release (Astagraf XL®) Once Daily vs Tacrolimus, Immediate Release BID; Logistic regression with occurrence of 5-point eGFR decline by Month 12 as response, with treatment group, planned Campath use, KDPI level (as recorded in IVRS), HLA Class II mismatch, recipient age, recipient gender, recipient race, and pre-transplant cPRA as fixed effects, and pooled site as a random effect with standard Variance Components covariance type; Test type: Superiority; p = 0.4995, Regression, Logistic; Odds Ratio (OR) = 1.212, 95% CI 2-sided [0.693 to 2.120]

19. Secondary Outcome: eGFR at Day 30, Day 90, Day 180, Day 270 and Day 365
Description: The eGFR was calculated using the MDRD formula.
Time Frame: Day 30, day 90, day 180, day 270 and day 365
Population: The mFAS consisted of all participants who were randomized and who received at least 1 dose of study drug (Astagraf XL or BID tacrolimus), and whose pretransplant cross-matched antibody samples did not demonstrate preformed DSA for the duration of the study. mFAS population with available data at each time point.
Measure: Mean (Standard Deviation); unit: mL/min/1.73 m^2
Arm/Group | Tacrolimus, Extended Release (Astagraf XL®) Once Daily | Tacrolimus, Immediate Release BID
Number analyzed (Participants) | 265 | 271
mL/min/1.73 m^2
  Day 30 | 50.86 (17.27) | 52.72 (19.40)
  Day 90: number analyzed (Participants) | 250 | 252
  Day 90 | 55.56 (16.00) | 57.10 (19.99)
  Day 180: number analyzed (Participants) | 230 | 229
  Day 180 | 56.81 (15.84) | 58.33 (17.51)
  Day 270: number analyzed (Participants) | 215 | 212
  Day 270 | 57.19 (16.84) | 59.04 (18.19)
  Day 365: number analyzed (Participants) | 204 | 193
  Day 365 | 58.25 (16.51) | 60.94 (17.83)

20. Secondary Outcome: Percentage of Participants With Graft Loss
Description: Graft loss was defined as re-transplantation, transplant nephrectomy, or a return to dialysis for at least a six week duration, or participants' death.
Time Frame: From date of transplant until 1 year
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Tacrolimus, Extended Release (Astagraf XL®) Once Daily | Tacrolimus, Immediate Release BID
Number analyzed (Participants) | 275 | 279
percentage of participants | 1.5 | 1.4

21. Secondary Outcome: Percentage of Participants Who Died
Description: Percentage of participants who died were reported.
Time Frame: From date of transplant until 1 year
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Tacrolimus, Extended Release (Astagraf XL®) Once Daily | Tacrolimus, Immediate Release BID
Number analyzed (Participants) | 275 | 279
percentage of participants | 0.7 | 0.7

22. Secondary Outcome: Percentage of Participants With Biopsy-Proven Acute Rejection (BPAR)
Description: Positivity was determined by local biopsy, central pathology, or reported adverse events.
Time Frame: From date of transplant until 1 year
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Tacrolimus, Extended Release (Astagraf XL®) Once Daily | Tacrolimus, Immediate Release BID
Number analyzed (Participants) | 275 | 279
percentage of participants | 7.6 | 8.2

23. Secondary Outcome: Percentage of Participants Who Were Lost to Follow-up
Description: Percentage of participants who were lost to follow-up were reported.
Time Frame: From date of transplant until 1 year
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Tacrolimus, Extended Release (Astagraf XL®) Once Daily | Tacrolimus, Immediate Release BID
Number analyzed (Participants) | 275 | 279
percentage of participants | 0 | 0.7

24. Secondary Outcome: Percentage of Participants With Either Graft Loss, Death, BPAR or Lost to Follow-up
Description: Percentage of participants with either graft loss, death, BPAR or lost to follow-up were reported.
Time Frame: From date of transplant until 1 year
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Tacrolimus, Extended Release (Astagraf XL®) Once Daily | Tacrolimus, Immediate Release BID
Number analyzed (Participants) | 275 | 279
percentage of participants | 9.1 | 10.4

25. Secondary Outcome: Percentage of Participants With Any Antibody-Mediated Rejection (ABMR)
Description: Percentage of participants with ABMR were reported. Central pathology reading was performed as per the 2007 Update to the Banff '97 classification. A positive assessment is defined as antibody mediated changes that are diagnosed as either acute ABMR or chronic active ABMR.
Time Frame: From date of transplant until month 14
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Tacrolimus, Extended Release (Astagraf XL®) Once Daily | Tacrolimus, Immediate Release BID
Number analyzed (Participants) | 275 | 279
percentage of participants | 1.6 | 0.7

26. Secondary Outcome: Percentage of Participants With Normal Biopsy Findings
Description: Percentage of participants with normal biopsy findings were reported.
Time Frame: From date of transplant until month 14
Population: The BAS consisted of all mFAS participants who had at least 1 post-transplant central pathology assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Tacrolimus, Extended Release (Astagraf XL®) Once Daily | Tacrolimus, Immediate Release BID
Number analyzed (Participants) | 123 | 136
percentage of participants | 6.5 | 4.4

27. Secondary Outcome: Percentage of Participants With C4d Deposition Without Active Rejection
Description: Percentage of participants with C4d deposition without active rejection were reported.
Time Frame: From date of transplant until month 14
Population: The BAS consisted of all mFAS participants who had at least 1 posttransplant central pathology assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Tacrolimus, Extended Release (Astagraf XL®) Once Daily | Tacrolimus, Immediate Release BID
Number analyzed (Participants) | 123 | 136
percentage of participants | 0.8 | 0.7

28. Secondary Outcome: Percentage of Participants With Acute ABMR
Description: Percentage of participants with acute ABMR were reported.
Time Frame: From date of transplant until month 14
Population: The BAS consisted of all mFAS participants who had at least 1 posttransplant central pathology assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Tacrolimus, Extended Release (Astagraf XL®) Once Daily | Tacrolimus, Immediate Release BID
Number analyzed (Participants) | 123 | 136
percentage of participants | 1.6 | 0.7

29. Secondary Outcome: Percentage of Participants With Grade I, II and III Acute ABMR
Description: Percentage of participants with grade I, II and III acute ABMR were reported. Central pathology reading was performed as per the 2007 Update to the Banff '97 classification. Acute ABMR was graded as Grade I: acute tubular necrosis-like -like minimal inflammation, Grade II: Capillary and or glomerular inflammation (ptc/g >0) and/or thromboses, and Grade III: arterial - v3.
Time Frame: From date of transplant until month 14
Population: The BAS consisted of all mFAS participants who had at least 1 post-transplant central pathology assessment. Only those BAS participants who had acute AMBR were included in the analyses.
Measure: Number; unit: percentage of participants
Arm/Group | Tacrolimus, Extended Release (Astagraf XL®) Once Daily | Tacrolimus, Immediate Release BID
Number analyzed (Participants) | 2 | 1
percentage of participants
  Grade I | 50 | 0
  Grade II | 50 | 100
  Grade III | 0 | 0

30. Secondary Outcome: Percentage of Participants With Chronic ABMR
Description: Percentage of participants with chronic ABMR were reported.
Time Frame: From date of transplant until month 14
Population: The BAS consisted of all mFAS participants who had at least 1 post-transplant central pathology assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Tacrolimus, Extended Release (Astagraf XL®) Once Daily | Tacrolimus, Immediate Release BID
Number analyzed (Participants) | 123 | 136
percentage of participants | 0 | 0

31. Secondary Outcome: Percentage of Participants With Borderline Changes
Description: Percentage of participants with borderline changes were reported.
Time Frame: From date of transplant until month 14
Population: The BAS consisted of all mFAS participants who had at least 1 post-transplant central pathology assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Tacrolimus, Extended Release (Astagraf XL®) Once Daily | Tacrolimus, Immediate Release BID
Number analyzed (Participants) | 123 | 136
percentage of participants | 14.6 | 14.7

32. Secondary Outcome: Percentage of Participants With Acute T-cell Mediated Rejection (TCMR)
Description: Percentage of participants with acute TCMR were reported.
Time Frame: From date of transplant until month 14
Population: The BAS consisted of all mFAS participants who had at least 1 post-transplant central pathology assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Tacrolimus, Extended Release (Astagraf XL®) Once Daily | Tacrolimus, Immediate Release BID
Number analyzed (Participants) | 123 | 136
percentage of participants | 6.5 | 5.9

33. Secondary Outcome: Percentage of Participants With Chronic TCMR
Description: Percentage of participants with chronic TCMR were reported.
Time Frame: From date of transplant until month 14
Population: The BAS consisted of all mFAS participants who had at least 1 post-transplant central pathology assessment. Only those BAS participants who had TCMR were included in the analyses.
Measure: Number; unit: percentage of participants
Arm/Group | Tacrolimus, Extended Release (Astagraf XL®) Once Daily | Tacrolimus, Immediate Release BID
Number analyzed (Participants) | 8 | 8
percentage of participants | 25 | 12.5

34. Secondary Outcome: Percentage of Participants With Grade I, II and III IFTA
Description: Percentage of participants with Grade I, II and III IFTA were reported. Central pathology reading was performed as per the 2007 Update to the Banff '97 classification. IFTA was graded as Grade I: mild interstitial fibrosis and tubular atrophy (<25% of cortical area), Grade II: moderate interstitial fibrosis and tubular atrophy (26-50% of cortical area), and Grade III: severe interstitial fibrosis and tubular atrophy/ loss (>50% of cortical area).
Time Frame: From date of transplant until month 14
Population: The BAS consisted of all mFAS participants who had at least 1 post-transplant central pathology assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Tacrolimus, Extended Release (Astagraf XL®) Once Daily | Tacrolimus, Immediate Release BID
Number analyzed (Participants) | 123 | 136
percentage of participants
  Grade I | 54.5 | 56.6
  Grade II | 18.7 | 15.4
  Grade III | 5.7 | 6.6

35. Secondary Outcome: Percentage of Participants With Any Additional Findings
Description: Percentage of participants with any additional findings (other than Normal biopsy, borderline changes, acute and chronic ABMR, Grade I, II, and III ABMR, C4D deposition, acute and chronic TCMR, Grade I, II, and III TCMR, Grade I, II and III IFTA, acute tubular necrosis, interstitial nephritis, pyelonephritis, bk virus, calcineurin inhibitor toxicity, hemolytic uremic syndrome and recurrent disease) were reported.
Time Frame: From date of transplant until month 14
Population: The BAS consisted of all mFAS participants who had at least 1 post-transplant central pathology assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Tacrolimus, Extended Release (Astagraf XL®) Once Daily | Tacrolimus, Immediate Release BID
Number analyzed (Participants) | 123 | 136
percentage of participants | 29.3 | 34.6

36. Secondary Outcome: Percentage of Participants With Glomerulitis (g) Biopsy Score Assessed Using Banff Lesion Scores
Description: Central pathology reading was performed as per the 2007 Update to the Banff '97 classification. Banff Lesion Scores assess the presence and the degree of histopathological changes in the different compartments of renal transplant biopsies, focusing primarily but not exclusively on the diagnostic features seen in rejection. [Roufosse C et. al 2018]. Here, Score 0= No glomerulitis, Score 1= <25% glomerulitis, Score 2= 25 to 75% glomerulitis and Score 3= >75% glomerulitis.
Time Frame: From date of transplant until month 14
Population: The BAS consisted of all mFAS participants who had at least 1 post-transplant central pathology assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Tacrolimus, Extended Release (Astagraf XL®) Once Daily | Tacrolimus, Immediate Release BID
Number analyzed (Participants) | 123 | 136
percentage of participants
  Banff Lesion Score 0 | 89.4 | 90.4
  Banff Lesion Score 1 | 5.7 | 6.6
  Banff Lesion Score 2 | 4.1 | 1.5
  Banff Lesion Score 3 | 0 | 0
  Not able to score | 0.8 | 1.5
Statistical Analysis 1: Comparison: Tacrolimus, Extended Release (Astagraf XL®) Once Daily vs Tacrolimus, Immediate Release BID; P-values obtained from the Exact Test of treatment arm by Banff scoring levels; Test type: Superiority; p = 0.6327, Fisher Exact

37. Secondary Outcome: Percentage of Participants With Tubulitis (t) Biopsy Score Assessed Using Banff Lesion Scores
Description: Central pathology reading was performed as per the 2007 Update to the Banff '97 classification. Banff Lesion Scores assess the presence and the degree of histopathological changes in the different compartments of renal transplant biopsies, focusing primarily but not exclusively on the diagnostic features seen in rejection. [Roufosse C et. al 2018]. Here, Score 0= No mononuclear cells in tubules or single focus of tubulitis only, Score 1= Foci with 1 to 4 mononuclear cells/tubular cross section (or 10 tubular cells), Score 2= Foci with 5 to 10 mononuclear cells/tubular cross section (or 10 tubular cells) and Score 3= Foci with >10 mononuclear cells/tubular cross section or the presence of ≥2 areas of tubular basement membrane destruction accompanied by i2/i3 inflammation and t2 elsewhere.
Time Frame: From date of transplant until month 14
Population: The BAS consisted of all mFAS participants who had at least 1 post-transplant central pathology assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Tacrolimus, Extended Release (Astagraf XL®) Once Daily | Tacrolimus, Immediate Release BID
Number analyzed (Participants) | 123 | 136
percentage of participants
  Banff Lesion Score 0 | 79.7 | 79.4
  Banff Lesion Score 1 | 16.3 | 15.4
  Banff Lesion Score 2 | 1.6 | 1.5
  Banff Lesion Score 3 | 1.6 | 2.9
  Not able to score | 0.8 | 0.7
Statistical Analysis 1: Comparison: Tacrolimus, Extended Release (Astagraf XL®) Once Daily vs Tacrolimus, Immediate Release BID; P-values obtained from the Exact Test of treatment arm by Banff scoring levels; Test type: Superiority; p = 0.9701, Fisher Exact

38. Secondary Outcome: Percentage of Participants With Intimal Arteritis (v) Biopsy Score Assessed Using Banff Lesion Scores
Description: Central pathology reading was performed as per the 2007 Update to the Banff '97 classification. Banff Lesion Scores assess the presence and the degree of histopathological changes in the different compartments of renal transplant biopsies, focusing primarily but not exclusively on the diagnostic features seen in rejection. [Roufosse C et. al 2018]. Here, Score 0= No arteritis, Score 1= Mild to moderate intimal arteritis in at least 1 arterial cross section, Score 2= Severe intimal arteritis with at least 25% luminal area lost in at least 1 arterial cross section and Score 3= Transmural arteritis and/or arterial fibrinoid change and medial smooth muscle necrosis with lymphocytic infiltrate in vessel.
Time Frame: From date of transplant until month 14
Population: The BAS consisted of all mFAS participants who had at least 1 post-transplant central pathology assessment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Tacrolimus, Extended Release (Astagraf XL®) Once Daily | Tacrolimus, Immediate Release BID
Number analyzed (Participants) | 123 | 136
Percentage of Participants
  Banff Lesion Score 0 | 93.5 | 94.9
  Banff Lesion Score 1 | 2.4 | 2.2
  Banff Lesion Score 2 | 2.4 | 0
  Banff Lesion Score 3 | 0 | 0
  Not able to score | 1.6 | 2.9
Statistical Analysis 1: Comparison: Tacrolimus, Extended Release (Astagraf XL®) Once Daily vs Tacrolimus, Immediate Release BID; P-values obtained from the Exact Test of treatment arm by Banff scoring levels; Test type: Superiority; p = 0.3127, Fisher Exact

39. Secondary Outcome: Percentage of Participants With Mononuclear Cell Interstitial Inflammation (i) Biopsy Score Assessed Using Banff Lesion Scores
Description: Central pathology reading was performed as per the 2007 Update to the Banff '97 classification. Banff Lesion Scores assess the presence and the degree of histopathological changes in the different compartments of renal transplant biopsies, focusing primarily but not exclusively on the diagnostic features seen in rejection. [Roufosse C et. al 2018]. Here, Score 0= No inflammation or in less than 10% of unscarred cortical parenchyma, Score 1= Inflammation in 10 to 25% of unscarred cortical parenchyma, Score 2= Inflammation in 26 to 50% of unscarred cortical parenchyma and Score 3= Inflammation in more than 50% of unscarred cortical parenchyma.
Time Frame: From date of transplant until month 14
Population: The BAS consisted of all mFAS participants who had at least 1 post-transplant central pathology assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Tacrolimus, Extended Release (Astagraf XL®) Once Daily | Tacrolimus, Immediate Release BID
Number analyzed (Participants) | 123 | 136
percentage of participants
  Banff Lesion Score 0 | 68.3 | 76.5
  Banff Lesion Score 1 | 26.8 | 17.6
  Banff Lesion Score 2 | 4.1 | 2.2
  Banff Lesion Score 3 | 0 | 2.9
  Not able to score | 0.8 | 0.7
Statistical Analysis 1: Comparison: Tacrolimus, Extended Release (Astagraf XL®) Once Daily vs Tacrolimus, Immediate Release BID; P-values obtained from the Exact Test of treatment arm by Banff scoring levels; Test type: Superiority; p = 0.0830, Fisher Exact

40. Secondary Outcome: Percentage of Participants With Glomerular Basement Membrane Double Contours (cg) Biopsy Score Assessed Using Banff Lesion Scores
Description: Central pathology reading was performed as per the 2007 Update to the Banff '97 classification. Banff Lesion Scores assess the presence and the degree of histopathological changes in the different compartments of renal transplant biopsies, focusing primarily but not exclusively on the diagnostic features seen in rejection. [Roufosse C et. al 2018]. Here, Score 0= No GBM double contours by light microscopy (LM) or electron microscopy (EM), Score 1= No GBM double contours by LM but GBM double contours (incomplete or circumferential) in at least 3 glomerular capillaries by EM or Double contours of the GBM in 1-25% of capillary loops in the most affected nonsclerotic glomerulus by LM , Score 2= Double contours affecting 26 to 50% of peripheral capillary loops in the most affected-glomerulus and Score 3= Double contours affecting more than 50% of peripheral capillary loops in the most affected-glomerulus.
Time Frame: From date of transplant until month 14
Population: The BAS consisted of all mFAS participants who had at least 1 post-transplant central pathology assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Tacrolimus, Extended Release (Astagraf XL®) Once Daily | Tacrolimus, Immediate Release BID
Number analyzed (Participants) | 123 | 136
percentage of participants
  Banff Lesion Score 0 | 93.5 | 93.4
  Banff Lesion Score 1 | 5.7 | 3.7
  Banff Lesion Score 2 | 0 | 1.5
  Banff Lesion Score 3 | 0 | 0
  Not able to score | 0.8 | 1.5
Statistical Analysis 1: Comparison: Tacrolimus, Extended Release (Astagraf XL®) Once Daily vs Tacrolimus, Immediate Release BID; P-values obtained from the Exact Test of treatment arm by Banff scoring levels; Test type: Superiority; p = 0.6022, Fisher Exact

41. Secondary Outcome: Percentage of Participants With Tubular Atrophy (ct) Biopsy Score Assessed Using Banff Lesion Scores
Description: Central pathology reading was performed as per the 2007 Update to the Banff '97 classification. Banff Lesion Scores assess the presence and the degree of histopathological changes in the different compartments of renal transplant biopsies, focusing primarily but not exclusively on the diagnostic features seen in rejection. [Roufosse C et. al 2018]. Here, Score 0= No tubular atrophy, Score 1= Tubular atrophy involving up to 25% of the area of cortical tubules, Score 2= Tubular atrophy involving 26 to 50% of the area of cortical tubules and Score 3= Tubular atrophy involving in >50% of the area of cortical tubules.
Time Frame: From date of transplant until month 14
Population: The BAS consisted of all mFAS participants who had at least 1 post-transplant central pathology assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Tacrolimus, Extended Release (Astagraf XL®) Once Daily | Tacrolimus, Immediate Release BID
Number analyzed (Participants) | 123 | 136
percentage of participants
  Banff Lesion Score 0 | 20.3 | 21.3
  Banff Lesion Score 1 | 53.7 | 55.9
  Banff Lesion Score 2 | 19.5 | 15.4
  Banff Lesion Score 3 | 5.7 | 6.6
  Not able to score | 0.8 | 0.7
Statistical Analysis 1: Comparison: Tacrolimus, Extended Release (Astagraf XL®) Once Daily vs Tacrolimus, Immediate Release BID; Test type: Superiority — P-values obtained from the Exact Test of treatment arm by Banff scoring levels; p = 0.9249, Fisher Exact

42. Secondary Outcome: Percentage of Participants With Interstitial Fibrosis (ci) Biopsy Score Assessed Using Banff Lesion Scores
Description: Central pathology reading was performed as per the 2007 Update to the Banff '97 classification. Banff Lesion Scores assess the presence and the degree of histopathological changes in the different compartments of renal transplant biopsies, focusing primarily but not exclusively on the diagnostic features seen in rejection. [Roufosse C et. al 2018]. Here, Score 0= Interstitial fibrosis in up to 5% of cortical area, Score 1= Interstitial fibrosis in 6 to 25%of cortical area (mild interstitial fibrosis), Score 2= Interstitial fibrosis in 26 to 50% of cortical area (moderate interstitial fibrosis) and Score 3= Interstitial fibrosis in >50% of cortical area (severe interstitial fibrosis).
Time Frame: From date of transplant until month 14
Population: The BAS consisted of all mFAS participants who had at least 1 post-transplant central pathology assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Tacrolimus, Extended Release (Astagraf XL®) Once Daily | Tacrolimus, Immediate Release BID
Number analyzed (Participants) | 123 | 136
percentage of participants
  Banff Lesion Score 0 | 21.1 | 20.6
  Banff Lesion Score 1 | 52.8 | 56.6
  Banff Lesion Score 2 | 19.5 | 15.4
  Banff Lesion Score 3 | 5.7 | 6.6
  Not able to score | 0.8 | 0.7
Statistical Analysis 1: Comparison: Tacrolimus, Extended Release (Astagraf XL®) Once Daily vs Tacrolimus, Immediate Release BID; P-values obtained from the Exact Test of treatment arm by Banff scoring levels; Test type: Superiority; p = 0.9136, Fisher Exact

43. Secondary Outcome: Percentage of Participants With Vascular Fibrous Intimal Thickening (cv) Biopsy Score Assessed Using Banff Lesion Scores
Description: Central pathology reading was performed as per the 2007 Update to the Banff '97 classification. Banff Lesion Scores assess the presence and the degree of histopathological changes in the different compartments of renal transplant biopsies, focusing primarily but not exclusively on the diagnostic features seen in rejection. [Roufosse C et. al 2018]. Here, Score 0= No chronic vascular changes, Score 1= Vascular narrowing of up to 25% luminal area by fibrointimal thickening, Score 2= Vascular narrowing of 26 to 50% luminal area by fibrointimal thickening and Score 3= Vascular narrowing of more than 50% luminal area by fibrointimal thickening.
Time Frame: From date of transplant until month 14
Population: The BAS consisted of all mFAS participants who had atleast 1 post-transplant central pathology assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Tacrolimus, Extended Release (Astagraf XL®) Once Daily | Tacrolimus, Immediate Release BID
Number analyzed (Participants) | 123 | 136
percentage of participants
  Banff Lesion Score 0 | 33.3 | 36
  Banff Lesion Score 1 | 40.7 | 41.2
  Banff Lesion Score 2 | 22 | 17.6
  Banff Lesion Score 3 | 2.4 | 2.2
  Not able to score | 1.6 | 2.9
Statistical Analysis 1: Comparison: Tacrolimus, Extended Release (Astagraf XL®) Once Daily vs Tacrolimus, Immediate Release BID; P-values obtained from the Exact Test of treatment arm by Banff scoring levels; Test type: Superiority; p = 0.8789, Fisher Exact

44. Secondary Outcome: Percentage of Participants With Arteriolar Hyalinosis (ah) Biopsy Score Assessed Using Banff Lesion Scores
Description: Central pathology reading was performed as per the 2007 Update to the Banff '97 classification. Banff Lesion Scores assess the presence and the degree of histopathological changes in the different compartments of renal transplant biopsies, focusing primarily but not exclusively on the diagnostic features seen in rejection. [Roufosse C et. al 2018]. Here, Score 0= No periodic acid-Schiff (PAS)-positive hyaline arteriolar thickening, Score 1= Mild to moderate PAS-positive hyaline thickening in at least 1 arteriole, Score 2= Moderate to severe PAS-positive hyaline thickening in more than 1 arteriole and Score 3= Severe PAS-positive hyaline thickening in many arterioles.
Time Frame: From date of transplant until month 14
Population: The BAS consisted of all mFAS participants who had at least 1 post-transplant central pathology assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Tacrolimus, Extended Release (Astagraf XL®) Once Daily | Tacrolimus, Immediate Release BID
Number analyzed (Participants) | 123 | 136
percentage of participants
  Banff Lesion Score 0 | 91.1 | 86.8
  Banff Lesion Score 1 | 4.1 | 5.9
  Banff Lesion Score 2 | 4.1 | 3.7
  Banff Lesion Score 3 | 0 | 2.2
  Not able to score | 0.8 | 1.5
Statistical Analysis 1: Comparison: Tacrolimus, Extended Release (Astagraf XL®) Once Daily vs Tacrolimus, Immediate Release BID; P-values obtained from the Exact Test of treatment arm by Banff scoring levels; Test type: Superiority; p = 0.5574, Fisher Exact

45. Secondary Outcome: Percentage of Participants With Peritubular Capillaritis (Ptc) Biopsy Score Assessed Using Banff Lesion Scores
Description: Central pathology reading was performed as per the 2007 Update to the Banff '97 classification. Banff Lesion Scores assess the presence and the degree of histopathological changes in the different compartments of renal transplant biopsies, focusing primarily but not exclusively on the diagnostic features seen in rejection. [Roufosse C et. al 2018]. Here, Score 0= Maximum number of leukocytes <3, Score 1= At least 1 leukocyte cell in ≥10% of cortical PTCs with 3-4 leukocytes in most severely involved PTC, Score 2= At least 1 leukocyte in ≥10% of cortical PTC with 5-10 leukocytes in most severely involved PTC and Score 3= At least 1 leukocyte in ≥10% of cortical PTC with >10 leukocytes in most severely involved PTC.
Time Frame: From date of transplant until month 14
Population: The BAS consisted of all mFAS participants who had at least 1 post-transplant central pathology assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Tacrolimus, Extended Release (Astagraf XL®) Once Daily | Tacrolimus, Immediate Release BID
Number analyzed (Participants) | 123 | 136
percentage of participants
  Banff Lesion Score 0 | 91.1 | 90.4
  Banff Lesion Score 1 | 3.3 | 5.1
  Banff Lesion Score 2 | 4.9 | 2.9
  Banff Lesion Score 3 | 0 | 0.7
  Not able to score | 0.8 | 0.7
Statistical Analysis 1: Comparison: Tacrolimus, Extended Release (Astagraf XL®) Once Daily vs Tacrolimus, Immediate Release BID; P-values obtained from the Exact Test of treatment arm by Banff scoring levels; Test type: Superiority; p = 0.8150, Fisher Exact

46. Secondary Outcome: Percentage of Participants With Mesangial Matrix Expansion (mm) Biopsy Score Assessed Using Banff Lesion Scores
Description: Central pathology reading was performed as per the 2007 Update to the Banff '97 classification. Banff Lesion Scores assess the presence and the degree of histopathological changes in the different compartments of renal transplant biopsies, focusing primarily but not exclusively on the diagnostic features seen in rejection. [Roufosse C et. al 2018]. Here, Score 0= No more than mild mesangial matrix increase in any glomerulus, Score 1= At least moderate mesangial matrix increase in up to 25% of nonsclerotic glomeruli, Score 2= At least moderate mesangial matrix increase in 26% to 50% of nonsclerotic glomeruli and Score 3= At least moderate mesangial matrix increase in >50% of nonsclerotic glomeruli.
Time Frame: From date of transplant until month 14
Population: The BAS consisted of all mFAS participants who had at least 1 post-transplant central pathology assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Tacrolimus, Extended Release (Astagraf XL®) Once Daily | Tacrolimus, Immediate Release BID
Number analyzed (Participants) | 123 | 136
percentage of participants
  Banff Lesion Score 0 | 87.8 | 91.2
  Banff Lesion Score 1 | 8.9 | 6.6
  Banff Lesion Score 2 | 2.4 | 0.7
  Banff Lesion Score 3 | 0 | 0
  Not able to score | 0.8 | 1.5
Statistical Analysis 1: Comparison: Tacrolimus, Extended Release (Astagraf XL®) Once Daily vs Tacrolimus, Immediate Release BID; P-values obtained from the Exact Test of treatment arm by Banff scoring levels; Test type: Superiority; p = 0.5673, Fisher Exact

47. Secondary Outcome: Time to First Occurrence of DSA
Description: as for outcome 4
Time Frame: From date of transplant until 1 year
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Tacrolimus, Extended Release (Astagraf XL®) Once Daily | Tacrolimus, Immediate Release BID
Number analyzed (Participants) | 275 | 279
days | NA (NA) — Analysis of data was not performed because it was not possible to define the exact date of occurrence since the data only recorded the date of sample collection which could not be interpreted as the date of first occurrence. | NA (NA) — Analysis of data was not performed because it was not possible to define the exact date of occurrence since the data only recorded the date of sample collection which could not be interpreted as the date of first occurrence.

48. Secondary Outcome: Time to First Occurrence of HLA-DQ DSA
Description: Time to first occurrence of HLA-DQ DSA was reported.
Time Frame: From date of transplant until 1 year
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Tacrolimus, Extended Release (Astagraf XL®) Once Daily | Tacrolimus, Immediate Release BID
Number analyzed (Participants) | 275 | 279
days | NA (NA) — Analysis of data was not performed because it was not possible to define the exact date of occurrence since the data only recorded the date of sample collection which could not be interpreted as the date of first occurrence. | NA (NA) — Analysis of data was not performed because it was not possible to define the exact date of occurrence since the data only recorded the date of sample collection which could not be interpreted as the date of first occurrence.

49. Secondary Outcome: Time to First Occurrence of C1q-binding DSA
Description: Time to first occurrence of C1q-binding DSA was reported.
Time Frame: From date of transplant until 1 year
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Tacrolimus, Extended Release (Astagraf XL®) Once Daily | Tacrolimus, Immediate Release BID
Number analyzed (Participants) | 275 | 279
days | NA (NA) — Analysis of data was not performed because it was not possible to define the exact date of occurrence since the data only recorded the date of sample collection which could not be interpreted as the date of first occurrence. | NA (NA) — Analysis of data was not performed because it was not possible to define the exact date of occurrence since the data only recorded the date of sample collection which could not be interpreted as the date of first occurrence.

50. Secondary Outcome: Time to First Occurrence of DSA IgG3 Isotype
Description: Time to first occurrence of DSA IgG3 isotype was reported.
Time Frame: From date of transplant until 1 year
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Tacrolimus, Extended Release (Astagraf XL®) Once Daily | Tacrolimus, Immediate Release BID
Number analyzed (Participants) | 275 | 279
days | NA (NA) — Analysis of data was not performed because it was not possible to define the exact date of occurrence since the data only recorded the date of sample collection which could not be interpreted as the date of first occurrence. | NA (NA) — Analysis of data was not performed because it was not possible to define the exact date of occurrence since the data only recorded the date of sample collection which could not be interpreted as the date of first occurrence.

51. Secondary Outcome: Time to First Occurrence of IA
Description: Time to first occurrence of IA was reported.
Time Frame: From date of transplant until 1 year
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Tacrolimus, Extended Release (Astagraf XL®) Once Daily | Tacrolimus, Immediate Release BID
Number analyzed (Participants) | 275 | 279
days | NA (NA) — Analysis of data was not performed because it was not possible to define the exact date of occurrence since the data only recorded the date of sample collection which could not be interpreted as the date of first occurrence. | NA (NA) — Analysis of data was not performed because it was not possible to define the exact date of occurrence since the data only recorded the date of sample collection which could not be interpreted as the date of first occurrence.

52. Secondary Outcome: Time to First Occurrence of TG on Biopsy
Description: Time to first occurrence of TG on biopsy was reported.
Time Frame: From date of transplant until 1 year
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Tacrolimus, Extended Release (Astagraf XL®) Once Daily | Tacrolimus, Immediate Release BID
Number analyzed (Participants) | 275 | 279
days | NA (NA) — Analysis of data was not performed because it was not possible to define the exact date of occurrence since the data only recorded the date of sample collection which could not be interpreted as the date of first occurrence. | NA (NA) — Analysis of data was not performed because it was not possible to define the exact date of occurrence since the data only recorded the date of sample collection which could not be interpreted as the date of first occurrence.

53. Secondary Outcome: Time to Occurrence of Death
Description: Time to occurrence of death was reported.
Time Frame: From date of transplant until 1 year
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Tacrolimus, Extended Release (Astagraf XL®) Once Daily | Tacrolimus, Immediate Release BID
Number analyzed (Participants) | 275 | 279
days | NA [NA to NA] — No data is reported since median and confidence interval was not estimable (that is, not reached) in either treatment group due to low number of events. | NA [NA to NA] — No data is reported since median and confidence interval was not estimable (that is, not reached) in either treatment group due to low number of events.

54. Secondary Outcome: Time to First Occurrence of Local BPAR
Description: Time to first occurrence of local BPAR was reported.
Time Frame: From date of transplant until 1 year
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Tacrolimus, Extended Release (Astagraf XL®) Once Daily | Tacrolimus, Immediate Release BID
Number analyzed (Participants) | 275 | 279
days | NA (NA) — Analysis of data was not performed because it was not possible to define the exact date of occurrence since the data only recorded the date of sample collection which could not be interpreted as the date of first occurrence. | NA (NA) — Analysis of data was not performed because it was not possible to define the exact date of occurrence since the data only recorded the date of sample collection which could not be interpreted as the date of first occurrence.

55. Secondary Outcome: Time to First Occurrence of Acute Forms of ABMR
Description: Time to first occurrence of acute forms of ABMR was reported.
Time Frame: From date of transplant until 1 year
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Tacrolimus, Extended Release (Astagraf XL®) Once Daily | Tacrolimus, Immediate Release BID
Number analyzed (Participants) | 275 | 279
days | NA (NA) — Analysis of data was not performed because it was not possible to define the exact date of occurrence since the data only recorded the date of sample collection which could not be interpreted as the date of first occurrence. | NA (NA) — Analysis of data was not performed because it was not possible to define the exact date of occurrence since the data only recorded the date of sample collection which could not be interpreted as the date of first occurrence.

56. Secondary Outcome: Time to First Occurrence of Chronic Forms of ABMR
Description: Time to first occurrence of chronic forms of ABMR was reported.
Time Frame: From date of transplant until 1 year
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Tacrolimus, Extended Release (Astagraf XL®) Once Daily | Tacrolimus, Immediate Release BID
Number analyzed (Participants) | 275 | 279
days | NA (NA) — Analysis of data was not performed because it was not possible to define the exact date of occurrence since the data only recorded the date of sample collection which could not be interpreted as the date of first occurrence. | NA (NA) — Analysis of data was not performed because it was not possible to define the exact date of occurrence since the data only recorded the date of sample collection which could not be interpreted as the date of first occurrence.

57. Secondary Outcome: Time to First Occurrence of Acute TCMR
Description: Time to first occurrence of acute TCMR was reported.
Time Frame: From date of transplant until 1 year
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Tacrolimus, Extended Release (Astagraf XL®) Once Daily | Tacrolimus, Immediate Release BID
Number analyzed (Participants) | 275 | 279
days | NA (NA) — Analysis of data was not performed because it was not possible to define the exact date of occurrence since the data only recorded the date of sample collection which could not be interpreted as the date of first occurrence. | NA (NA) — Analysis of data was not performed because it was not possible to define the exact date of occurrence since the data only recorded the date of sample collection which could not be interpreted as the date of first occurrence.

58. Secondary Outcome: Time to First Occurrence of Chronic TCMR
Description: Time to first occurrence of chronic TCMR was reported.
Time Frame: From date of transplant until 1 year
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Tacrolimus, Extended Release (Astagraf XL®) Once Daily | Tacrolimus, Immediate Release BID
Number analyzed (Participants) | 275 | 279
days | NA (NA) — Analysis of data was not performed because it was not possible to define the exact date of occurrence since the data only recorded the date of sample collection which could not be interpreted as the date of first occurrence. | NA (NA) — Analysis of data was not performed because it was not possible to define the exact date of occurrence since the data only recorded the date of sample collection which could not be interpreted as the date of first occurrence.

59. Secondary Outcome: Time to First Occurrence of Borderline Changes
Description: Time to first occurrence of borderline changes was reported.
Time Frame: From date of transplant until 1 year
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Tacrolimus, Extended Release (Astagraf XL®) Once Daily | Tacrolimus, Immediate Release BID
Number analyzed (Participants) | 275 | 279
days | NA (NA) — Analysis of data was not performed because it was not possible to define the exact date of occurrence since the data only recorded the date of sample collection which could not be interpreted as the date of first occurrence. | NA (NA) — Analysis of data was not performed because it was not possible to define the exact date of occurrence since the data only recorded the date of sample collection which could not be interpreted as the date of first occurrence.

60. Secondary Outcome: Time to First Occurrence of IFTA
Description: Time to first occurrence of IFTA was reported.
Time Frame: From date of transplant until 1 year
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Tacrolimus, Extended Release (Astagraf XL®) Once Daily | Tacrolimus, Immediate Release BID
Number analyzed (Participants) | 275 | 279
days | NA (NA) — Analysis of data was not performed because it was not possible to define the exact date of occurrence since the data only recorded the date of sample collection which could not be interpreted as the date of first occurrence. | NA (NA) — Analysis of data was not performed because it was not possible to define the exact date of occurrence since the data only recorded the date of sample collection which could not be interpreted as the date of first occurrence.

61. Secondary Outcome: Percentage of Participants With Treatment-emergent Adverse Event(TEAEs), Related TEAEs, Treatment-emergent Serious Adverse Event (TESAEs), Related TESAEs, TEAEs Leading to Discontinuation of Study Treatment and TEAEs Leading to Death
Description: A TEAE was defined as an Adverse Event (AE) observed on or after the day of starting the administration of the test drug/comparative drug.
Time Frame: From first dose of study drug up to 7 days after last dose of study drug (up to 2 years)
Population: The Safety Analysis Set (SAF) consisted of all participants who enrolled into the study and took at least 1 dose of study medication and was used for all safety, tolerability, and medication compliance related variables.
Measure: Number; unit: percentage of participants
Arm/Group | Tacrolimus, Extended Release (Astagraf XL®) Once Daily | Tacrolimus, Immediate Release BID
Number analyzed (Participants) | 288 | 287
percentage of participants
  TEAEs | 99.7 | 98.6
  TEAEs related to study treatment | 77.8 | 70.7
  TESAEs | 56.6 | 47.4
  TESAEs related to study treatment | 27.4 | 23.7
  TEAEs causing discontinuation of study treatment | 16.3 | 13.9
  TEAEs leading to death | 0.7 | 0.7

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 7 days after last dose of study drug (up to 2 years)
Description: The SAF consisted of all participants who enrolled into the study and took at least 1 dose of study medication and was used for all safety, tolerability, and medication compliance related variables.
Arm/Group | Tacrolimus, Extended Release (Astagraf XL®) Once Daily | Tacrolimus, Immediate Release BID
All-Cause Mortality (participants affected / at risk) | 2/288 | 2/287
Serious Adverse Events (participants affected / at risk) | 163/288 | 136/287
Other Adverse Events (participants affected / at risk) | 285/288 | 278/287
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tacrolimus, Extended Release (Astagraf XL®) Once Daily (N=288) | Tacrolimus, Immediate Release BID (N=287)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 6 (6)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 3 (4)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Methaemoglobinaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 5 (7) | 2 (2)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 3 (3) | 2 (3)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Aortic valve stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 2 (2)
Bradycardia (Cardiac disorders) | 3 (3) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 2 (2) | 0 (0)
Left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Pulseless electrical activity (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 2 (2)
Congenital cystic kidney disease (Congenital, familial and genetic disorders) | 0 (0) | 2 (2)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hyperparathyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Hyperparathyroidism tertiary (Endocrine disorders) | 2 (2) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 6 (10)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Diabetic gastroparesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 7 (7) | 11 (11)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gastrointestinal necrosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 4 (4)
Impaired gastric emptying (Gastrointestinal disorders) | 2 (5) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intra-abdominal fluid collection (Gastrointestinal disorders) | 2 (2) | 3 (3)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (6) | 5 (6)
Obstructive pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Odynophagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 3 (3) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (2) | 0 (0)
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (2)
Vomiting (Gastrointestinal disorders) | 4 (7) | 7 (10)
Asthenia (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 2 (2) | 5 (5)
Death (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0)
Haemorrhagic cyst (General disorders) | 1 (1) | 0 (0)
Implant site extravasation (General disorders) | 1 (1) | 0 (0)
Incarcerated hernia (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 1 (1)
Peripheral swelling (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 9 (10) | 8 (11)
Biliary tract disorder (Hepatobiliary disorders) | 1 (1) | 0 (0)
Gallbladder necrosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatitis alcoholic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0)
Kidney transplant rejection (Immune system disorders) | 12 (13) | 14 (17)
Renal transplant failure (Immune system disorders) | 0 (0) | 1 (1)
Transplant rejection (Immune system disorders) | 2 (2) | 2 (2)
Abdominal abscess (Infections and infestations) | 0 (0) | 1 (1)
Abscess neck (Infections and infestations) | 0 (0) | 1 (1)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1)
Arteriovenous fistula site infection (Infections and infestations) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 4 (4) | 4 (4)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 4 (6) | 4 (6)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 2 (2) | 6 (6)
Coccidioidomycosis (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 2 (2)
Cytomegalovirus colitis (Infections and infestations) | 0 (0) | 1 (1)
Cytomegalovirus infection (Infections and infestations) | 3 (3) | 2 (2)
Cytomegalovirus viraemia (Infections and infestations) | 4 (4) | 6 (6)
Diabetic foot infection (Infections and infestations) | 1 (1) | 0 (0)
Disseminated cytomegaloviral infection (Infections and infestations) | 0 (0) | 1 (1)
Enterobacter bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Enterococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Enterococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Enterovirus infection (Infections and infestations) | 1 (1) | 0 (0)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 1 (2)
Escherichia infection (Infections and infestations) | 0 (0) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 3 (4) | 2 (3)
Fungaemia (Infections and infestations) | 0 (0) | 1 (1)
Fungal oesophagitis (Infections and infestations) | 1 (1) | 0 (0)
Gangrene (Infections and infestations) | 0 (0) | 2 (2)
Gastroenteritis (Infections and infestations) | 3 (3) | 3 (3)
Gastroenteritis norovirus (Infections and infestations) | 2 (2) | 2 (2)
Gastroenteritis viral (Infections and infestations) | 4 (4) | 1 (1)
Incision site abscess (Infections and infestations) | 0 (0) | 2 (3)
Infected cyst (Infections and infestations) | 1 (1) | 1 (1)
Infection in an immunocompromised host (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 1 (1)
Klebsiella bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 2 (2) | 0 (0)
Lower respiratory tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1)
Lymph node tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Necrotising soft tissue infection (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 3 (4) | 2 (2)
Paronychia (Infections and infestations) | 1 (1) | 0 (0)
Perirectal abscess (Infections and infestations) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0)
Peritonitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 10 (11) | 7 (8)
Pneumonia klebsiella (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia legionella (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia pseudomonal (Infections and infestations) | 1 (1) | 0 (0)
Polyomavirus-associated nephropathy (Infections and infestations) | 1 (1) | 1 (1)
Pseudomonal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 2 (2)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 2 (2)
Rhinovirus infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 7 (7) | 10 (10)
Septic shock (Infections and infestations) | 1 (1) | 2 (2)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 3 (4)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Streptococcal urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2)
Urinary tract infection (Infections and infestations) | 16 (17) | 11 (12)
Urinary tract infection bacterial (Infections and infestations) | 2 (2) | 2 (2)
Urinary tract infection enterococcal (Infections and infestations) | 2 (2) | 2 (2)
Urosepsis (Infections and infestations) | 1 (1) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Viral pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Vulval abscess (Infections and infestations) | 0 (0) | 1 (1)
Vulval cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 1 (1) | 1 (1)
Wound infection staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Delayed graft function (Injury, poisoning and procedural complications) | 5 (5) | 4 (4)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Graft complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incision site pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Perirenal haematoma (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Post procedural haematuria (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Psychosis postoperative (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Transplant dysfunction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ureteric anastomosis complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Wound haematoma (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 10 (12) | 8 (9)
Blood potassium increased (Investigations) | 1 (1) | 0 (0)
Clostridium test positive (Investigations) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0)
Histology abnormal (Investigations) | 1 (1) | 0 (0)
Immunosuppressant drug level increased (Investigations) | 0 (0) | 1 (1)
Mycobacterium test positive (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 5 (7)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 7 (7) | 2 (2)
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 15 (16) | 5 (6)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Lactic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteitis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Post transplant lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Carotid artery occlusion (Nervous system disorders) | 0 (0) | 1 (1)
Central nervous system haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Central nervous system lesion (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Hypertensive encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Myelopathy (Nervous system disorders) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1)
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Status epilepticus (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 2 (2) | 3 (3)
Device dislocation (Product Issues) | 0 (0) | 1 (1)
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 2 (2) | 2 (3)
Acute kidney injury (Renal and urinary disorders) | 26 (33) | 31 (36)
Azotaemia (Renal and urinary disorders) | 2 (2) | 0 (0)
Bladder outlet obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Focal segmental glomerulosclerosis (Renal and urinary disorders) | 2 (3) | 0 (0)
Haematuria (Renal and urinary disorders) | 2 (2) | 2 (2)
Haemorrhage urinary tract (Renal and urinary disorders) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 3 (3) | 5 (6)
Perinephric collection (Renal and urinary disorders) | 3 (4) | 5 (5)
Renal artery stenosis (Renal and urinary disorders) | 2 (2) | 1 (1)
Renal artery thrombosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal pain (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal tubular injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal tubular necrosis (Renal and urinary disorders) | 2 (2) | 1 (1)
Renal vein thrombosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 (0) | 1 (1)
Ureteric obstruction (Renal and urinary disorders) | 2 (2) | 0 (0)
Ureteric stenosis (Renal and urinary disorders) | 1 (1) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinoma (Renal and urinary disorders) | 0 (0) | 2 (2)
Acquired phimosis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Scrotal oedema (Reproductive system and breast disorders) | 0 (0) | 1 (2)
Testicular swelling (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Nasal necrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin necrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Swelling face (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Therapy change (Surgical and medical procedures) | 1 (1) | 0 (0)
Arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0)
Arteriovenous fistula (Vascular disorders) | 0 (0) | 1 (1)
Axillary vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 6 (6) | 5 (5)
Extremity necrosis (Vascular disorders) | 2 (2) | 1 (1)
Extrinsic iliac vein compression (Vascular disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 2 (2)
Haemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 5 (5) | 4 (4)
Hypertensive crisis (Vascular disorders) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 2 (2) | 4 (4)
Ischaemia (Vascular disorders) | 0 (0) | 1 (1)
Lymphocele (Vascular disorders) | 2 (2) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 2 (2)
Steal syndrome (Vascular disorders) | 1 (1) | 1 (1)
Subclavian vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Thrombophlebitis superficial (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tacrolimus, Extended Release (Astagraf XL®) Once Daily (N=288) | Tacrolimus, Immediate Release BID (N=287)
Anaemia (Blood and lymphatic system disorders) | 42 (46) | 37 (45)
Leukocytosis (Blood and lymphatic system disorders) | 12 (12) | 21 (23)
Leukopenia (Blood and lymphatic system disorders) | 66 (74) | 58 (67)
Neutropenia (Blood and lymphatic system disorders) | 20 (23) | 28 (30)
Thrombocytopenia (Blood and lymphatic system disorders) | 14 (14) | 18 (18)
Tachycardia (Cardiac disorders) | 27 (28) | 24 (25)
Abdominal distension (Gastrointestinal disorders) | 14 (15) | 21 (27)
Abdominal pain (Gastrointestinal disorders) | 31 (34) | 35 (39)
Constipation (Gastrointestinal disorders) | 90 (101) | 100 (113)
Diarrhoea (Gastrointestinal disorders) | 128 (165) | 115 (160)
Dyspepsia (Gastrointestinal disorders) | 24 (26) | 24 (29)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 15 (18) | 9 (9)
Nausea (Gastrointestinal disorders) | 101 (131) | 104 (133)
Vomiting (Gastrointestinal disorders) | 41 (54) | 61 (77)
Asthenia (General disorders) | 21 (23) | 14 (15)
Chest pain (General disorders) | 15 (15) | 12 (12)
Fatigue (General disorders) | 45 (48) | 45 (51)
Oedema (General disorders) | 10 (12) | 17 (18)
Oedema peripheral (General disorders) | 53 (63) | 53 (64)
Pyrexia (General disorders) | 28 (37) | 38 (44)
BK virus infection (Infections and infestations) | 45 (47) | 37 (37)
Cytomegalovirus viraemia (Infections and infestations) | 18 (21) | 15 (15)
Nasopharyngitis (Infections and infestations) | 21 (23) | 17 (19)
Upper respiratory tract infection (Infections and infestations) | 25 (27) | 31 (32)
Urinary tract infection (Infections and infestations) | 50 (65) | 44 (77)
Delayed graft function (Injury, poisoning and procedural complications) | 15 (15) | 30 (30)
Incision site pain (Injury, poisoning and procedural complications) | 24 (25) | 47 (50)
Procedural pain (Injury, poisoning and procedural complications) | 55 (62) | 91 (105)
Blood creatinine increased (Investigations) | 37 (40) | 43 (49)
Viral test positive (Investigations) | 10 (11) | 18 (18)
Weight increased (Investigations) | 16 (18) | 14 (14)
Decreased appetite (Metabolism and nutrition disorders) | 12 (14) | 20 (20)
Dehydration (Metabolism and nutrition disorders) | 14 (14) | 21 (23)
Diabetes mellitus (Metabolism and nutrition disorders) | 18 (19) | 19 (19)
Hypercalcaemia (Metabolism and nutrition disorders) | 14 (15) | 18 (18)
Hyperglycaemia (Metabolism and nutrition disorders) | 37 (41) | 58 (62)
Hyperkalaemia (Metabolism and nutrition disorders) | 81 (106) | 79 (102)
Hyperphosphataemia (Metabolism and nutrition disorders) | 18 (20) | 21 (22)
Hypocalcaemia (Metabolism and nutrition disorders) | 37 (43) | 41 (42)
Hypoglycaemia (Metabolism and nutrition disorders) | 12 (14) | 16 (20)
Hypokalaemia (Metabolism and nutrition disorders) | 38 (39) | 37 (44)
Hypomagnesaemia (Metabolism and nutrition disorders) | 124 (142) | 124 (143)
Hyponatraemia (Metabolism and nutrition disorders) | 19 (21) | 18 (18)
Hypophosphataemia (Metabolism and nutrition disorders) | 122 (133) | 122 (133)
Metabolic acidosis (Metabolism and nutrition disorders) | 50 (57) | 60 (70)
Vitamin D deficiency (Metabolism and nutrition disorders) | 38 (38) | 35 (35)
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 (18) | 16 (22)
Back pain (Musculoskeletal and connective tissue disorders) | 19 (20) | 17 (17)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 12 (12) | 21 (22)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 17 (20) | 23 (27)
Dizziness (Nervous system disorders) | 34 (41) | 30 (36)
Headache (Nervous system disorders) | 46 (58) | 38 (43)
Tremor (Nervous system disorders) | 94 (99) | 84 (89)
Anxiety (Psychiatric disorders) | 12 (14) | 24 (29)
Insomnia (Psychiatric disorders) | 40 (42) | 44 (47)
Dysuria (Renal and urinary disorders) | 27 (30) | 21 (23)
Haematuria (Renal and urinary disorders) | 25 (26) | 30 (30)
Proteinuria (Renal and urinary disorders) | 5 (5) | 15 (15)
Urinary retention (Renal and urinary disorders) | 13 (14) | 18 (18)
Cough (Respiratory, thoracic and mediastinal disorders) | 26 (26) | 20 (22)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 32 (34) | 30 (38)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 23 (27) | 21 (22)
Alopecia (Skin and subcutaneous tissue disorders) | 24 (24) | 15 (15)
Pruritus (Skin and subcutaneous tissue disorders) | 18 (18) | 21 (23)
Hypertension (Vascular disorders) | 53 (57) | 50 (53)
Hypotension (Vascular disorders) | 41 (44) | 45 (51)
Orthostatic hypotension (Vascular disorders) | 13 (14) | 19 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript prior to publication for review and comment as specified in the Investigator Agreement.

DOCUMENTS (2):
  • Study Protocol (2018-05-25): https://cdn.clinicaltrials.gov/large-docs/91/NCT02723591/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-09): https://cdn.clinicaltrials.gov/large-docs/91/NCT02723591/SAP_001.pdf